CLINICAL TRIAL: NCT02461238
Title: Etude Fruits et Légumes à la Maison (FLAM)
Brief Title: Impact of Vouchers and Nutrition Education on the Consumption of Fruits and Vegetables Among Vulnerable Families (FLAM)
Acronym: FLAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Paris 13 (Other)
Collaborators: Direction Générale de la Santé, France (Other); Maison de la Santé de la ville de Saint Denis (Unknown); Ville de Saint Denis (Unknown); Programme Malin (Unknown); Institut National de Prévention et d'Education pour la Sante (Unknown)
Responsible Party: Principal Investigator, Serge HERCBERG, Head of department, University of Paris 13
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UParis13
Record Dates: First submitted 2015-05-27; First posted 2015-06-03 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Primary Prevention; Nutrition Policy
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vouchers (Active Comparator): Families included in the Voucher arm will receive vouchers for fruits and vegetables by mail every month for a period of 1 year coupled to nutritional education from a dietician
  Interventions: Other: Vouchers; Other: Nutrition education
- Control (Other): Families included in the control arm will only receive nutritional education
  Interventions: Other: Nutrition education

INTERVENTIONS:
Other: Vouchers — The vouchers sent to families can be used in supermarkets for fresh, frozen or canned fruits and vegetables, excluding potatoes. The amount of the vouchers takes into account family composition, calculated to correspond to a serving per day per person.
  Arms: Vouchers
Other: Nutrition education — Nutrition education workshops taught by a dietician

SUMMARY:
The purpose of this study is to assess whether fruit and vegetables vouchers combined with educational support may increase fruits and vegetables consumption of children aged 3 to 10 living in vulnerable families in Saint-Denis, France.

ELIGIBILITY:
Inclusion Criteria:

* At least one of the following criteria :

  * One or both parent(s) is/are beneficiary of resource allocation condition
  * One or both parent is/are unemployed
  * Household income below the poverty line
* Minimum of one child aged 3 to 10 at the time of the inclusion
* Stable housing

Exclusion Criteria:

* Parent is under 18
* Family having no permanent address or planned move within a year
* Consent form unsigned
* Opposition of a parent for their child's inclusion in the study
* Higher household income of 1700 euros per month for single-parent family or higher than 2 000 euros for other families

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Proportion of small consumers of fruits and vegetables among children | 12 months
  Average daily intake of fruits and vegetables is measured using a food frequency questionnaire, in order to determine the proportion of small consumer of fruits and vegetables. Before-after comparisons will be made in each arm, and compared between both arms at T+1.
  Subjects consuming less than 3.5 servings of fruit and vegetables per day are defined as small consumers.

SECONDARY OUTCOMES:
Proportion of small consumers of fruits and vegetables among adults (parents) | 12 months
  Average daily intake of fruits and vegetables is measured using a food frequency questionnaire, in order to determine the proportion of small consumer of fruits and vegetables. Before-after comparisons will be made in each arm, and compared between both arms at T+1.
  Subjects consuming less than 3.5 servings of fruit and vegetables per day are defined as small consumers.
Utilization rate of vouchers (voucher arm) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maison de la Santé, Saint-Denis, France

REFERENCES:
- [Derived] Buscail C, Gendreau J, Daval P, Lombrail P, Hercberg S, Latino-Martel P, Julia C. Impact of fruits and vegetables vouchers on food insecurity in disadvantaged families from a Paris suburb. BMC Nutr. 2019 Apr 4;5:26. doi: 10.1186/s40795-019-0289-4. eCollection 2019. PMID 32153939
- [Derived] Buscail C, Margat A, Miszkowicz T, Gendreau J, Daval P, Lombrail P, Hercberg S, Latino-Martel P, Maurice A, Julia C. Recruitment of precarious families in an interventional study: Lessons from the French "Fruits and vegetables at home" (FLAM) trial. Contemp Clin Trials Commun. 2018 Nov 2;12:161-168. doi: 10.1016/j.conctc.2018.10.008. eCollection 2018 Dec. PMID 30480163
- [Derived] Buscail C, Margat A, Petit S, Gendreau J, Daval P, Lombrail P, Hercberg S, Latino-Martel P, Maurice A, Julia C. Fruits and vegetables at home (FLAM): a randomized controlled trial of the impact of fruits and vegetables vouchers in children from low-income families in an urban district of France. BMC Public Health. 2018 Aug 28;18(1):1065. doi: 10.1186/s12889-018-5908-5. PMID 30153820